CLINICAL TRIAL: NCT01895881
Title: Estrogen Therapy as Prevention in the Progression of Aneurysm
Brief Title: Estrogen Therapy as Prevention in the Progression of Aneurysm (EPPA) Trial
Acronym: EPPA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to Recruit Participants
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Michael Chen, M.D., Associate Professor of Neurology, Neurosurgery and Radiology, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EPPA - 12101906
Record Dates: First submitted 2013-05-24; First posted 2013-07-11 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Cerebral Aneurysm; Menopause; Treatment
Keywords: Intracranial Aneurysm; Estradiol
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Estradiol Daily (Experimental): 1 mg Estradiol daily for 180 days.
  Interventions: Drug: Estradiol
- Placebo (Placebo Comparator): Placebo for 180 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Estradiol
  Arms: Estradiol Daily
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study aims to determine if hormone replacement therapy, given during perimenopause may prevent the progression of saccular cerebral aneurysms.

DETAILED DESCRIPTION:
This is a prospective, randomized, placebo-control trial to test the effect of estradiol in the prevention of progression of cerebral aneurysms. To evaluate the effect, each subject will be treated with either oral estradiol or placebo for 6 months. Subjects will be randomly assigned to 1 of 2 groups as follows:

Double Blind Treatment Group Open-Label Regimen A1 1 mg Estradiol daily for 180 days B1 Placebo for 180 days

Each group will be given oral Progesterone (3300 mg) for 10 days at the end of 90 days regardless of menstrual pattern. Subjects will be asked to keep a menstrual calendar throughout the trial. Serum markers will be drawn at baseline and every 90 days with the results blinded until the end of the trial. Magnetic resonance angiography (MRA) studies of the brain will be performed at month 6.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy women, 40-52 years of age.
* At least one documented saccular intracranial cerebral aneurysm detected via catheter angiography, magnetic resonance angiography or computed tomography angiography.
* Clinical diagnosis of perimenopause, defined as regular or irregular menses with or without vasomotor symptoms.

Exclusion Criteria:

* Known or suspected estrogen-dependent neoplasia.
* Endometrial proliferation, hyperplasia, or malignancy at screening.
* Known hypersensitivity to estrogens, progestins.
* History of myocardial infarction, ischemic heart disease, lipid disorder, or congestive heart failure.
* Known or suspected pregnancy, or recent breast feeding (within 6 months).

Ages: 40 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Effect of low dose estradiol on a panel of serum markers. | Change in levels of serum markers from baseline and six months.
  Parallel design double-blind placebo controlled trial to assess the effect of low dose estradiol on serum lipoprotein (a), serum elastase, and homocysteine.

SECONDARY OUTCOMES:
Radiographic change in the cerebral vasculature after treatment. | From date of randomization to six months.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chen, MD, Principal Investigator — Rush University Medical Center; Barbara Soltes, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chen M, Ouyang B, Goldstein-Smith L, Feldman L. Oral contraceptive and hormone replacement therapy in women with cerebral aneurysms. J Neurointerv Surg. 2011 Jun;3(2):163-6. doi: 10.1136/jnis.2010.003855. Epub 2010 Dec 17. PMID 21990811
- [Result] Ding C, Toll V, Ouyang B, Chen M. Younger age of menopause in women with cerebral aneurysms. J Neurointerv Surg. 2013 Jul;5(4):327-31. doi: 10.1136/neurintsurg-2012-010364. Epub 2012 Jun 13. PMID 22700728